CLINICAL TRIAL: NCT03489083
Title: Heat-induced Extracellular HSP72 Release is Blunted in Elderly Diabetic People in Comparison With Healthy Middle-aged and Older Adults But is Partially Restored by Strength Training
Brief Title: Heat Shock Response is Blunted in Elderly Diabetic People But Recovered by Strength Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Maurício Krause, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UFRGS 1.614.907
Record Dates: First submitted 2018-03-20; First posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-03

CONDITIONS: Type 2 Diabetes Mellitus; Aging
Keywords: Diabetes; Heat Shock Response; Aging; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The aim of this study was to compare the heat shock response (HSR) between healthy middle-aged adults (45-59 years old), healthy elderly adults (> 60 y.o.) and type 2 diabetic elderly people (> 60 y.o.). In addition, considering the effects of strength exercise in promoting health, we aimed to test the effects of strength training over the HSR in diabetic elderly people.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trained Group (Experimental): Subjects performing strength training three times per week for twelve weeks.
  Interventions: Other: Strength training
- No Training Group (Placebo Comparator): Subjects performing "placebo" stretching/relaxing session once a week (for adherence purposes) for twelve weeks.
  Interventions: Other: No Training

INTERVENTIONS:
Other: Strength training — Strength training was performed three times per week for twelve weeks. Supervised (by qualified sport and exercise scientists) exercise was performed in a gym on three non-consecutive days of the week. Each session lasted ~60 min and consisted of a warm up, the resistance exercise training and a cool down. The training programme consisted of a combination of upper and lower body exercises using gym equipments, free weights and body weight as the primary resistance. The twelve weeks of strength training were divided into three mesocycles of four weeks each. The resistance training was performed using two to three sets per exercise at intensities between 12-15 repetition maximum-RM.
  Arms: Trained Group
Other: No Training — Control group performed a "placebo" stretching/relaxing session once a week (for adherence purposes) for twelve weeks. To avoid any significant adaptation, all stretching exercises (for large muscle groups only) were performed at very low intensity without any significant discomfort.
  Arms: No Training Group

SUMMARY:
The aim of this study was to compare the heat shock response (HSR) between healthy middle-aged adults, healthy elderly adults and type 2 diabetic elderly people. In addition, considering the effects of strength exercise in promoting health, we aimed to test the effects of strength training over the HSR in diabetic elderly people. Thirty (19 females and 11 males) sedentary non-smoking participants volunteered for this study (11 healthy middle-age adults, 7 healthy old adults and 12 diabetic old subjects, previously diagnosed by their personal physicians).

Firstly, venous blood samples were obtained from all participants to test the HSR. They were divided in three groups: healthy middle-age adults (45-59 y.o.), healthy elderly adults and elderly diabetic (> 60 y.o.). As we identify that diabetic people presented a poor HSR, we submit the diabetic group to a twelve-week resistance exercise training to verify if this intervention could improve the HS response.

Diabetic subjects were randomly (1:1 block randomization) allocated in one of the two groups: Trained and Control (no training). Strength training was performed three times per week while the control group performed a "placebo" stretching/relaxing session once a week (for adherence purposes). Both interventions had twelve weeks of duration. To avoid any significant adaptation, all stretching exercises (for large muscle groups only) were performed at very low intensity without any significant discomfort.

Supervised (by qualified sport and exercise scientists) exercise was performed in a gym on three non-consecutive days of the week. Each session lasted ~60 min and consisted of a warm up, the resistance exercise training and a cool down. The training programme consisted of a combination of upper and lower body exercises using gym equipments, free weights and body weight as the primary resistance. The twelve weeks of strength training were divided into three mesocycles of four weeks each. Exercises included leg press, knee extensions and leg curls, biceps curls, triceps extensions, lat pull-downs, shoulder press, bench press and abdominal crunch. Before the start of the training period, subjects completed a familiarization session to practice the exercises they would further perform during the training sessions, where the exercise load was individually tested. The resistance training was performed using two to three sets per exercise at intensities between 12-15 repetition maximum-RM.

ELIGIBILITY:
Inclusion Criteria:

* . Inclusion criteria for diabetic people were HbA1c ≤ 7,5% (within the last six months), controlled blood pressure and no use of insulin.

Exclusion Criteria:

* Participants were excluded if they reported a history of myocardial infarction, cardiac illness, vascular disease, stroke, major systemic disease or any condition that would prevent them from engaging in an exercise study; or if they were already engaging in two or more planned and structured exercise sessions per week (in the last six months).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Heat Shock Response Change. | Before and After twelve weeks of exercise training.
  Capacity of cells to express and export heat shock protein 72kDa in response to heat (ng/mL).

SECONDARY OUTCOMES:
hs-CRP Change. | Before and After twelve weeks of exercise training.
  Marker of Inflammation measured in mg/L.
Body composition Change. | Before and After twelve weeks of exercise training.
  Body mass index (in Kg/m2).
TNF-a Change. | Before and After twelve weeks of exercise training.
  Marker of Inflammation measured in pg/mL.
IL-10 Change. | Before and After twelve weeks of exercise training.
  Marker of Inflammation measured in pg/mL.
Visceral Adipose Tissue Change. | Before and After twelve weeks of exercise training.
  Amount of visceral adipose tissue measured in millimeters (mm).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All data, including HSR, body composition, inflammatory and oxidative stress markers and metabolites.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After training completion
Access Criteria: All volunteers